CLINICAL TRIAL: NCT06684184
Title: Safety and Efficacy of Blinatumomab in Refractory Myasthenia Gravis
Brief Title: Blinatumomab in Refractory Myasthenia Gravis (BLINA-MG)
Acronym: BLINA-MG
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Zhongming Qiu (Other)
Responsible Party: Sponsor-Investigator, Zhongming Qiu, Professor, Xinqiao Hospital of Chongqing
Organization: Xinqiao Hospital of Chongqing (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-254-01
Record Dates: First submitted 2024-10-16; First posted 2024-11-12 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Myasthaenia Gravis
MeSH Terms: interventions — blinatumomab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment group (Experimental)
  Interventions: Drug: Blinatumomab

INTERVENTIONS:
Drug: Blinatumomab — The initial dose is 9 µ g, administered intravenously continuously for 5 days, with a total dose of 38.5 µ g. After stopping the medication for one week, the patient received a second infusion of Blinatumomab for a total of 5 days, with a total dose of 38.5 µ g.

SUMMARY:
The goal of this clinical trial is to evaluating the efficacy and safety of Blinatumomab in the treatment of refractory myasthenia gravis and exploring the immunological mechanisms of Blinatumomab therapy in refractory myasthenia gravis. The main questions it aims to answer are:

Will Blinatumomab improve the symptoms of participants? What medical problems do participants have when using Blinatumomab?

Participants will:

Continuous intravenous infusion of Blinatumomab for 5 days, pause for one week, and continue continuous intravenous infusion for 5 days Visit the clinic once every 1 month for checkups and tests Keep a diary of their symptoms

ELIGIBILITY:
Inclusion Criteria:

* 18 years old ≤ Age ≤ 75 years old
* patients with a Myasthenia Gravis Activities of Daily Living (MG-ADL) scale score of 6 or higher, and an ocular muscle score constituting less than 50% of the total score
* after receiving an adequate course of at least two conventional immunotherapeutic drugs (including both steroidal and non-steroidal immunosuppressants), the Post-Intervention Status (PIS) remains unchanged or worsens; or after receiving an adequate course of at least two conventional immunotherapeutic drugs, the PIS improves, but the MG-ADL score is still ≥6 points and persists for at least half a year; or after receiving an adequate course of at least two conventional immunotherapeutic drugs, the PIS is in remission or improvement, yet during the regular tapering of immunotherapeutic drugs, there are still at least two annual exacerbations of disease symptoms (MG-ADL score ≥6 points); or after the occurrence of a crisis, despite multiple immunotherapies such as intravenous immunoglobulin, plasmapheresis, and high-dose intravenous methylprednisolone, and active infection control, the patient still cannot be weaned off the ventilator due to MG-induced respiratory muscle weakness for more than 14 days
* positive for anti-AChR, and/or anti-MuSK, and/or anti-LRP4 antibodies.
* patient or their legal representative signs an informed consent form in writing

Exclusion Criteria:

* pregnant or lactating women
* individuals with an allergy to Blinatumomab
* individuals who have undergone thymectomy within the 12 months prior to baseline or who are planning to have a thymectomy during the 12-week study period
* individuals who have received biologic agents targeting CD19 or CD20 within 6 months prior to baseline are eligible for enrollment (subjects with CD19 or CD20 positive B cell counts above the lower limit of normal are allowed to participate)
* within the 3 months prior to baseline, use of Ecuzumab and Tocilizumab
* received intravenous immunoglobulin or plasma exchange therapy within 4 weeks prior to baseline
* currently participating in other clinical studies

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-11-30 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Myasthenia Gravis Activities of Daily Living (MG-ADL) Scale | At the 12th week
  The minimum value is 0, and maximum value is 24. higher scores mean a worse outcome. The primary endpoint is the proportion of patients who achieved a reduction of at least 2 points in the MG-ADL score by week 12 and did not undergo rescue therapy.

IPD SHARING:
Plan to Share IPD: No